CLINICAL TRIAL: NCT01829074
Title: Predictive Value of Subjective and Objective Measurement Tools for Extraesophageal Reflux
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Respiratory Technology Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 13RT001
Record Dates: First submitted 2013-04-02; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Laryngopharyngeal Reflux
Keywords: Laryngopharyngeal Reflux; Hoarseness; Throat Clearing; Globus Sensation
MeSH Terms: conditions — Laryngopharyngeal Reflux; Hoarseness; Globus Sensation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Acid reflux can cause many symptoms in the throat, including discomfort or pain, and difficulty with breathing and voice problems. Doctors have different ways of diagnosing and treating the reflux that causes these symptoms, and they are trying to better understand what the best ways are to treat the patients with these symptoms.

Usually, a doctor will prescribe medication for reflux based on the symptoms a patient complains of. Sometimes it works and the patient gets better, sometimes it does not work and the patient's condition does not improve. The doctor will also use findings from an examination with an endoscope in the patient's throat to see if there is any damage that might have been caused by reflux. One new device that doctors use to help them diagnose reflux has a sensor on the end of a tube that goes through the nose and rests in the throat. This sensor measures the acid reflux for 24 hours, showing the doctor when acid reflux occurs.

The study doctors are performing this research study to help them understand more about acid reflux disease, and the best ways to diagnose and treat their patients who have acid reflux.

The study involves procedures, medications and devices that are already used regularly in doctors' offices and hospitals. The experimental part of this research is blinding the study doctor to the results of the pH study until the end of a three month course of antireflux medication, and performing a second pH study to measure change in acid exposure.

Hypothesis: The Restech pH study helps identify patients who will respond positively to acid inhibitory therapy, and patients whose study normalizes will have better Symptomatic response rates than those whose pH levels fail to normalize.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the ENT clinic for distressing symptoms of hoarseness, laryngitis, and/or recurrent throat clearing for at least 3 months duration. Determined not to be caused by another factor, such as allergies or poor vocal hygiene.
* Laryngoscopic examination performed on day of enrollment
* Indications present for a 24 hour oropharyngeal pH study (Restech)
* Indication to begin a 3 month course of antireflux therapy (Figure 1) based on symptom presentation and widely accepted otolaryngologic findings
* Willing to return to clinic in 3 months for follow up pH study
* Willing to participate in weekly phone calls with the study investigator to discuss compliance with medication and lifestyle modifications.

Exclusion Criteria:

* Expected non-compliance with the equipment and/or instructions (according the protocol) given by the investigator.
* Any subjects with significant medical conditions that, in the investigator's judgment, would compromise the subject's health and safety.
* Subjects who have undergone previous antireflux surgery
* Subjects treated for reflux, either with Proton Pump Inhibitors (PPI's) or H2RAs in the past 4 weeks
* Subjects previously treated for reflux, either with antireflux medication or surgery
* Subjects with alternative work schedules affecting nighttime sleep periods (i.e. nighttime shift employees)
* Subjects with conditions that contraindicate use of PPIs, as listed on product labeling.
* Women who are pregnant, or nursing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Otolaryngology practices of the co-investigators with certain symptoms consistent with Laryngopharyngeal reflux: hoarseness, globus sensation, and/or recurrent throat clearing for more than 3 months
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Symptomatic Improvement (treatment result) in the group of patients who are "LPR negative" (normal pH study) at baseline versus the symptomatic improvement of the patients who are "LPR positive" (abnormal pH study) at baseline. | 12/2013 (up to 8 months)
  After their first set of visits, the patients will be followed during their 3 month course of anti-reflux medications (PPIs). After three months, the patients will be asked to repeat the VAS and validated symptoms questionnaires. These will be compared to their baseline scores to measure symptomatic improvement.
  Using the criterion of 50% improvement in symptoms as the cutoff point (dividing factor), the two populations will be divided further into two groups: responders and non-responders.
  The amount of responders in each group will be compared to see if there is a greater proportion of responders in the group of patients who were LPR positive at baseline than in the group who were LPR negative at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nimish Vakil, MD, Principal Investigator — University of Wisconsin, Madison, USA